CLINICAL TRIAL: NCT06760026
Title: Cosmetic Results With Tissue Adhesive (2-octylcyanoacrylate) vs. Subdermal Sutures in Cesarean Section: Single-blind Randomized Clinical Trial
Brief Title: Cosmetic Results With Tissue Adhesive vs. Subdermal Sutures in Cesarean Section
Acronym: ADTID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ricardo A Gutierrez Ramirez, MD, MSc, FACOG (Other)
Responsible Party: Sponsor-Investigator, Ricardo A Gutierrez Ramirez, MD, MSc, FACOG, Titular professor, Universidad Nacional Autonoma de Honduras
Organization: Universidad Nacional Autonoma de Honduras (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PGO-UNAH-48-4-2025
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Cesarean Wound Repair; Cesarean Section Scar; Cosmetic Appearance of Cesarean Scar; Tissue Adhesives
Keywords: Cesarean Wound Repair; Cesarean section scar; cosmetic appearance of cesarean scar; tissue adhesives

STUDY DESIGN:
Intervention Model Description: Single-blind, parallel-group, randomized clinical trial of superiority
Who Masked: Outcomes Assessor
Masking Description: Both the patient and the principal investigator will know the intervention, the data analyst researcher does not know the group to which the patients have been assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): use 2-octyl cyanoacrylate tissue adhesive applied continuously over the Pfannenstiel-type cesarean incision
  Interventions: Procedure: 2-octyl cyanoacrylate tissue adhesive applied continuously over the Pfannenstiel-type cesarean incision
- Control (Active Comparator): wound closure with subdermal sutures using 2-0 nylon thread
  Interventions: Procedure: subdermal suture

INTERVENTIONS:
Procedure: 2-octyl cyanoacrylate tissue adhesive applied continuously over the Pfannenstiel-type cesarean incision — 2-octyl cyanoacrylate tissue adhesive applied continuously over the Pfannenstiel-type cesarean incision
  Arms: Intervention
Procedure: subdermal suture — wound closure with subdermal sutures using 2-0 nylon thread, under the same evaluation scheme
  Arms: Control

SUMMARY:
Morbidity associated with post-cesarean wound closure, including cosmetically unfavorable scarring, is a significant concern in obstetrics, impacting patient satisfaction and recovery. Recent advances have introduced the use of tissue adhesives, such as 2-octylcyanoacrylate, which promise to improve cosmetic outcomes and reduce postoperative complications. This study will evaluate different tissue adhesive application schedules, keeping the total dose constant, to determine whether the method of application influences cosmetic results and the incidence of postoperative complications

DETAILED DESCRIPTION:
In Honduras, as in many parts of the world, cesarean section is a common obstetric practice. The choice of wound closure method in this procedure has significant implications not only in terms of the patient's physical health, but also in her psychological and aesthetic well-being. The scar resulting from a cesarean section can have a lasting impact on a woman's perception of her own body, affecting her self-esteem and quality of life.

Historically, in Honduras, the use of subdermal sutures with nylon thread has been preferred for the closure of post-cesarean section wounds. However, with advances in medical technology, tissue adhesives have emerged as a promising alternative, potentially offering a better cosmetic outcome, faster application, and more comfortable recovery for the patient.

This study is crucial in the Honduran context for several reasons:

1. improved Cosmetic Outcomes and Patient Satisfaction: By comparing two methods of wound closure, this study seeks to identify the technique that offers better cosmetic results, which could significantly improve the satisfaction and psychological well-being of patients undergoing elective cesarean sections.
2. Adaptation to Local Resources: In a country like Honduras, where health resources may be limited, it is essential to optimize the use of technologies and surgical materials. This study will provide valuable information on the feasibility and efficacy of tissue adhesives compared to the traditional method, taking into account factors such as cost and availability of materials.
3. Reduction of Postoperative Complications: By evaluating and comparing the incidence of complications associated with each closure method, the study could contribute to improve surgical practices and reduce the incidence of postoperative complications, which is of great relevance in the context of public health in Honduras.
4. Impact on Resource Management in the Health System: In the context of a country with possibly limited health resources such as Honduras, it is essential to evaluate not only the clinical efficacy of surgical techniques, but also their cost-effectiveness. This study will provide information on the relative costs of the use of tissue adhesives compared to subdermal sutures, which is relevant for planning and resource allocation in the health system.
5. Fostering Research and Evidence-Based Medicine in Honduras: This study will contribute to the growing need for contextualized medical research in Honduras, promoting the practice of evidence-based medicine that takes into account local realities and the specific needs of the population.

Objective: To evaluate the effects on morbidity and postoperative cosmetic outcomes of the use of tissue adhesive versus subdermal sutures in Pfannenstiel-type cesarean sections.

ELIGIBILITY:
Inclusion Criteria:

* Submission of a signed and dated informed consent form.
* Declared willingness to comply with all study procedures and availability for the duration of the study.
* Pregnant patient at 37 or more weeks gestation, scheduled for elective cesarean section at the Hospital Materno Infantil.
* Cesarean section performed in the Maternity and Children's Hospital, operating room.
* Literate patient, able to understand and respond to the study questions, with body mass index less than 30.
* Possess cell phone or other means of communication to facilitate postoperative follow-up.
* Residing in the city of Tegucigalpa, Honduras, to ensure accessibility to scheduled follow-up visits.

Exclusion Criteria:

* Patients under 18 years of age.
* Patients with diagnosed psychiatric illnesses that may interfere with their ability to give informed consent or follow the study protocol.
* Pregnant patients with complications that may affect the healing process or increase the risk of postoperative complications, such as severe preeclampsia.
* Diabetes.
* Collagen diseases.
* Autoimmune diseases (rheumatoid arthritis, Crohn's disease).
* Vascular diseases (vasculitis).
* Coagulation disorders (thrombophilia).
* Pregnant patients with premature rupture of membranes, since this may influence the choice of timing and method of cesarean section.
* Pregnant patients diagnosed with chorioamnionitis, which represents an increased risk of postoperative infection.
* Pregnant patients diagnosed with acute abdomen, which may require emergency surgical management that is not compatible with standard cesarean section procedures.
* Pregnant patients with multiple pregnancies, since this could complicate the cesarean section procedure and affect the results of the study.
* Presence of major fetal malformations that may require additional interventions at birth.
* Fetal stillbirth

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the OSAS Scale score | One month from the first intervention until 6 months
  The OSAS score is based on the assessment of several aspects of a scar, and each of these aspects is scored individually. Each variable uses a 10-point scoring system, where 1 represents normal foot. The scores of the individual variables can be added together to obtain a total score ranging from 5 to 50, where 5 represents normal skin.
  Items typically assessed include:
  * Vascularity: Refers to the presence of visible blood vessels or red coloration in the scar.
  * Pigmentation: Assesses whether the scar has a different color than the surrounding skin.
  * Thickness: Refers to the height or prominence of the scar above the level of the surrounding skin.
  * Relief: Assesses the texture of the scar compared to the surrounding skin.
  * Flexibility: Measures how stiff or flexible the scar is compared to the surrounding skin.

SECONDARY OUTCOMES:
PSAS scale score | One month from the first intervention until 6 months
  The Patient Scar Assessment Scale (PSAS) consists of 6 items on scar-related pain, itching, color, stiffness, thickness, and irregularity. Each item uses a 10-point scoring system, summed to give a total score ranging from 6 to 60, where 6 represents normal skin with no associated symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A. Gutierrez Ramirez, MD, MSc, Study Director — Universidad Nacional Autonoma de Honduras
Locations (1):
- Hospital Escuela, Tegucigalpa, Francisco Morazán Department, Honduras

IPD SHARING:
Plan to Share IPD: No
It is not necessary, none of the 18 HIPAA identifiers will be placed

REFERENCES:
- [Background] Cromi A, Ghezzi F, Gottardi A, Cherubino M, Uccella S, Valdatta L. Cosmetic outcomes of various skin closure methods following cesarean delivery: a randomized trial. Am J Obstet Gynecol. 2010 Jul;203(1):36.e1-8. doi: 10.1016/j.ajog.2010.02.001. Epub 2010 Apr 24. PMID 20417924